CLINICAL TRIAL: NCT05571358
Title: Virtual Reality to Improve Low-back Pain and Pelvic Pain During Pregnancy for a Multicentre Randomized Controlled Trial
Brief Title: Virtual Reality to Improve Low-back Pain and Pelvic Pain During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Francisco Jose García Lopez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR - LBP
Record Dates: First submitted 2022-06-23; First posted 2022-10-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain; Pelvic Pain
MeSH Terms: conditions — Low Back Pain; Pelvic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Following clinical practice guidelines, subjects in the control group will receive multidisciplinary rehabilitation programmes with coordinated delivery of supervised exercise therapy, cognitive behavioural therapy (education on pain), as well as therapeutic massage to relieve low back pain during pregnancy.
- Virtual Reality (Nature Trek) (Experimental): * Subjects in the experimental group will receive the same treatment described for the control group.
  * Subjects in the experimental group will receive an additional Virtual Reality Intervention (VRi).
  Interventions: Device: Virtual Reality (Nature Trek)

INTERVENTIONS:
Device: Virtual Reality (Nature Trek) — At the end of each session, participants will experience an immersive virtual landscape displayed by Nature Trek VR software (httpp://naturetreksvr.com/). First, participants will be placed in a sit down position and guided for their breathing control during 5 minutes ("meditation Lotus option"). After that, they will be encouraged to freely move around a relaxing virtual environment during 15 minutes taking special attention to soothing sounds of nature. The themes environment will be selected based on the preferences of the participants.
  At the beginning of the study, advice is given on general care, in physical activity and issues concerning drug intake. Patients are advised to refrain from any other specific training during the intervention period. Any deviations from the adherence and practice of the VRi are recorded daily, noting any adverse incidents.
  Arms: Virtual Reality (Nature Trek)

SUMMARY:
A large percentage of women suffer low back and pelvic pain both during and after pregnancy. There are several factors to which these complaints are attributed, even affecting their daily lives. It is identified that many of these women do not receive adequate health care, however, different physiotherapeutic interventions are recommended to alleviate these conditions, presenting moderate levels of evidence. Virtual reality (VR) is presented as a complementary and promising treatment method to physiotherapy for the improvement of fundamental variables such as perceived pain and pain avoidance. The main objective is to evaluate the efficacy of a combined VR and physiotherapy program of 4 weeks duration compared to a standard physiotherapy intervention in pregnant women with low back pain and pelvic pain for the improvement of pain avoidance, pain intensity, disability and functional level. As a secondary objective the investigators propose to investigate patient satisfaction with the VR intervention. This research will be carried out by means of a multicenter randomized controlled clinical trial in pregnant patients residing in the provinces of Seville and Malaga with a diagnosis of low back pain and pelvic pain during pregnancy. The alternative hypothesis of this research is that the implementation of a Virtual Reality program together with standard physiotherapy in pregnant patients with low back and pelvic pain presents better clinical results obtained with the current standard intervention, which may represent an opportunity to define new policies and interventions for these pathologies and their consequences.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman over 18 years old
* Pregnant woman with Low Back Pain, Pelvic Pain (PP) or both conditions with symptomatic character.
* Pregnant woman between the 12th and 36th week of gestation, corresponding to the 2nd and 3rd trimester.
* Pain intensity greater than 4/10 on VAS, indicating moderate-severe pain.
* Live in Sevilla or Malaga during the research period.

Exclusion Criteria:

* Patients with LBP or PP pain prior to pregnancy.
* Cognitive ability not suitable for the use of technological tools.
* Patients with absolute or relative contraindications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Fear-Avoidance Components Scale (FACS) | Baseline FACS
  FACS. Pain-related fear avoidance (FA), a common problem for patients with painful medical conditions, involves pain-related catastrophizing cognitions, hypervigilance, and avoidance behaviors, which can ultimately lead to decreased functioning, depression, and disability. (FACS) was developed, which incorporates important components of previous FA- related measures, and includes components of the FA model not previously considered in the earlier-developed questionnaires. The FACS has 20 items, each measured on a 6-point Likert scale, for total possible score of 100 and the lowest possible score of 0, requesting the respondent to either: (5) completely agree; (4) mostly agree; (3) slightly agree; (2) slightly disagree; (1) mostly disagree; (0) completely disagree. Higher scores are intended to indicate higher levels of FA.
The Fear-Avoidance Components Scale (FACS) | 4 weeks FACS
  FACS. Pain-related fear avoidance (FA), a common problem for patients with painful medical conditions, involves pain-related catastrophizing cognitions, hypervigilance, and avoidance behaviors, which can ultimately lead to decreased functioning, depression, and disability. (FACS) was developed, which incorporates important components of previous FA- related measures, and includes components of the FA model not previously considered in the earlier-developed questionnaires. The FACS has 20 items, each measured on a 6-point Likert scale, for total possible score of 100 and the lowest possible score of 0, requesting the respondent to either: (5) completely agree; (4) mostly agree; (3) slightly agree; (2) slightly disagree; (1) mostly disagree; (0) completely disagree. Higher scores are intended to indicate higher levels of FA.
Pain Intensity | Baseline
  The Visual Analog Scale (VAS) has been used in previous studies investigating changes in pain and, specifically, in all the randomized trials of interventions for back pain in pregnancy included in or published since the Cochrane and systematic reviews. The VAS was used for assessment of pain before and after the intervention. Measurement will be performed with a 10-cm scale marked with 1-cm increments. Pain felt by participants will be recorded. Pain was rated on a scale of 0 a 10, with 10 representing the most excruciating pain. The value indicated on the scale by the participants was used as the score.
Pain Intensity | 4 weeks
  The Visual Analog Scale (VAS) has been used in previous studies investigating changes in pain and, specifically, in all the randomized trials of interventions for back pain in pregnancy included in or published since the Cochrane and systematic reviews. The VAS was used for assessment of pain before and after the intervention. Measurement will be performed with a 10-cm scale marked with 1-cm increments. Pain felt by participants will be recorded. Pain was rated on a scale of 0 a 10, with 10 representing the most excruciating pain. The value indicated on the scale by the participants was used as the score.
Disability and Physical function | Baseline RMDQ
  The investigators focus on the 2 back-specific measures of function recommended in the "core-set," the Roland-Morris disability Questionnaire (RMDQ) and the Oswestry Disability Index (ODI). The RMDQ will be used for measurement of the severity of disability in participants who had less severe Low Back Pain (LBP). There are 24 categories comprised of yes or no questions. Each participant can have a maximum score of 24. Scoring closer to 24 indicates greater functional disability.
Disability and Physical function | 4 weeks RMDQ
  The investigators focus on the 2 back-specific measures of function recommended in the "core-set," the Roland-Morris disability Questionnaire (RMDQ) and the Oswestry Disability Index (ODI). The RMDQ will be used for measurement of the severity of disability in participants who had less severe Low Back Pain (LBP). There are 24 categories comprised of yes or no questions. Each participant can have a maximum score of 24. Scoring closer to 24 indicates greater functional disability.
Disability and Physical function | Baseline ODI
  The investigators focus on the 2 back-specific measures of function recommended in the "core-set," the Roland-Morris disability Questionnaire (RMDQ) and the Oswestry Disability Index (ODI). The Oswestry low-back pain disability index (ODI) will be completed by the participants and included 10 questions assessing activities of daily living in order to examine the functional level when experiencing LBP. Each category will be scored from zero to five with regard to the severity of disability caused during daily life.
Disability and Physical function | 4 weeks ODI
  The investigators focus on the 2 back-specific measures of function recommended in the "core-set," the Roland-Morris disability Questionnaire (RMDQ) and the Oswestry Disability Index (ODI). The Oswestry low-back pain disability index (ODI) will be completed by the participants and included 10 questions assessing activities of daily living in order to examine the functional level when experiencing LBP. Each category will be scored from zero to five with regard to the severity of disability caused during daily life.

SECONDARY OUTCOMES:
Satisfaction with Virtual Reality intervention | Baseline USEQ
  The User Satisfaction Evaluation Questionnaire (USEQ) is a questionnaire that is designed to properly evaluate the satisfaction of the user (which constitutes part of usability) in virtual rehabilitation systems. The USEQ questionnaire is composed of the set of questions in the SEQ that evaluate satisfaction. The USEQ has six questions with a five-point Likert Scale. The total score of the USEQ questionnaire ranges from 6 (poor satisfaction) to 30 (excellent satisfaction). To calculate this total score, we consider all of the questions to be positive, except for Q5, which is considered to be a negative question. The numerical value of the positive questions is used to calculate the score (for instance, if the patient selects 4 in Q1, then 4 is added to the total score). The negative question subtracts the numerical value of the response from 6 and then adds this result to the total score (for instance, if the patient selects 2 in Q5, then 4 is added to the total score).
Satisfaction with Virtual Reality intervention | 4 weeks USEQ
  To assess the Satisfaction with the Virtual Rehabilitation Systems the investigators will use the User Satisfaction Evaluation Questionnaire (USEQ). The USEQ is a questionnaire that is designed to properly evaluate the satisfaction of the user (which constitutes part of usability) in virtual rehabilitation systems. The USEQ questionnaire is composed of the set of questions in the SEQ that evaluate satisfaction. The USEQ has six questions with a five-point Likert Scale. The total score of the USEQ questionnaire ranges from 6 (poor satisfaction) to 30 (excellent satisfaction).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Lopez FJ, Pastora-Bernal JM, Moreno-Morales N, Estebanez-Perez MJ, Linan-Gonzalez A, Martin-Valero R. Virtual reality to improve low-back pain and pelvic pain during pregnancy: a pilot RCT for a multicenter randomized controlled trial. Front Med (Lausanne). 2023 Sep 4;10:1206799. doi: 10.3389/fmed.2023.1206799. eCollection 2023. PMID 37731709

DOCUMENTS (1):
  • Study Protocol (2022-06-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT05571358/Prot_000.pdf